CLINICAL TRIAL: NCT06683391
Title: Updating pReventive and Treatment guidelinEs for Mild hypOglycemia in Individuals Living With Type 1 Diabetes During the erA of Continuous gLucose Monitoring: The REMODAL Trial
Brief Title: Updating Preventive and Treatment Guidelines for Hypoglycemia in Individuals Living With Type 1 Diabetes
Acronym: REMODAL
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Institut de Recherches Cliniques de Montreal (Other)
Responsible Party: Principal Investigator, Rémi Rabasa-Lhoret, Vice President clinic and clinical research, Professor, Institut de Recherches Cliniques de Montreal
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 2025-1295
Record Dates: First submitted 2024-11-06; First posted 2024-11-12 (Actual); Last update posted 2025-02-25 (Actual); Status verified 2025-02

CONDITIONS: Type 1 Diabetes
Keywords: type 1 diabetes; hypoglycemia
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Hypoglycemia | interventions — Carbohydrates; Organization and Administration; Therapeutics

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Masking Description: open-label masking
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- 16g CHO at < 4.0 mmol/L (Reactive Approach) (Placebo Comparator): Participants receive 16 grams of carbohydrate only when their CGM reading falls below 4.0 mmol/L, in line with the traditional "reactive" approach. This arm serves as a control, reflecting current hypoglycemia treatment guidelines, allowing comparison to proactive interventions.
  Interventions: Behavioral: Oral Carbohydrate (CHO) Administration for Hypoglycemia Prevention and Treatment
- 8g CHO at 5.0 mmol/L (Proactive Approach) (Experimental): Participants receive 8 grams of carbohydrate when their CGM reading reaches a proactive threshold of 5.0 mmol/L. This arm tests whether a lower amount of CHO, administered at a higher glucose level, can effectively prevent hypoglycemia with minimal caloric intake.
  Interventions: Behavioral: Oral Carbohydrate (CHO) Administration for Hypoglycemia Prevention and Treatment
- 16g CHO at 5.0 mmol/L (Proactive Approach) (Experimental): Participants receive 16 grams of carbohydrate at the proactive threshold of 5.0 mmol/L. This arm examines if a slightly higher dose of CHO at the same proactive threshold provides additional preventive benefits compared to 8 grams, while still aiming to avoid hypoglycemia and limit subsequent glucose fluctuations.
  Interventions: Behavioral: Oral Carbohydrate (CHO) Administration for Hypoglycemia Prevention and Treatment

INTERVENTIONS:
Behavioral: Oral Carbohydrate (CHO) Administration for Hypoglycemia Prevention and Treatment — The intervention in the REMODAL trial involves administering specific amounts of oral carbohydrates (CHO) at different glucose thresholds to evaluate the effectiveness of proactive versus reactive hypoglycemia management strategies in adults with Type 1 diabetes using continuous glucose monitoring (CGM). Participants will undergo three distinct interventions, each designed to test a different amount and timing of CHO intake.

SUMMARY:
The REMODAL trial is a randomized crossover study aiming to update treatment guidelines for mild hypoglycemia in people with Type 1 diabetes using continuous glucose monitoring (CGM) technology. The study will assess whether treating mild hypoglycemia proactively (at a glucose threshold of 5.0 mmol/L) with lower doses of carbohydrate (CHO) is more effective than the traditional reactive approach (treatment at < 4.0 mmol/L). The goal is to reduce hypoglycemia frequency and improve quality of life, while minimizing caloric intake and rebound hyperglycemia.

DETAILED DESCRIPTION:
The REMODAL trial explores an individualized, proactive approach to treat mild hypoglycemia in individuals with Type 1 diabetes (T1D) who use CGM. Traditional guidelines, established in the 1980s, recommend the "15g/15min rule" - consuming 15g of CHO every 15 minutes for glucose levels below 4.0 mmol/L. However, these guidelines may no longer be optimal with the advancements in insulin therapies and CGM, which provide real-time glucose data and predict glucose trends.

In this study, 32 adult participants with T1D will receive three interventions to test different amounts and timing of CHO intake under real-life conditions. These are as follows:

1. 8g of CHO at a threshold of 5.0 mmol/L (proactive approach).
2. 16g of CHO at a threshold of 5.0 mmol/L (proactive approach).
3. 16g of CHO at a threshold of < 4.0 mmol/L (traditional reactive approach).

The primary outcome is the prevention rate of hypoglycemic episodes under each intervention, with additional measures on glucose levels, time spent in hypoglycemia, and rebound hyperglycemia. The study also considers differences in glucose management between multiple daily injections, continuous subcutaneous insulin infusion, and automated insulin delivery systems, which may affect CHO needs. This study hopes to redefine effective hypoglycemia management in the modern era of diabetes care, providing personalized recommendations to improve glycemic control and overall quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 years and older
* Clinical diagnosis of Type 1 diabetes for at least 1 year
* Currently treated with multiple daily insulin injections (MDI), continuous subcutaneous insulin infusion (CSII), or automated insulin delivery (AID) systems
* HbA1c level below 9.0%
* Equal distribution of male and female participants, as well as MDI/CSII and AID users

Exclusion Criteria:

* Gastroparesis
* Significant cardiac rhythm abnormalities
* Clinically significant microvascular complications such as nephropathy (eGFR < 40 ml/min) or severe proliferative retinopathy
* Diagnosis of epilepsy
* Pregnancy or currently breastfeeding
* Severe hypoglycemic episode within 1 month prior to inclusion
* Macrovascular events or uncorrected hypokalemia (K+ < 3.5 mmol/L) within 3 months prior to inclusion
* Anticipated treatment changes during the trial period
* Inability to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Self-representation of gender identity
Enrollment: 32 (Estimated)
Dates: Start 2025-02-06 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Percentage of Hypoglycemia Prevention with 16g CHO at 5.0 mmol/L | 60 minutes
  The primary outcome will measure the percentage of hypoglycemic episodes prevented when participants consume 16 grams of carbohydrate (CHO) at a proactive threshold of 5.0 mmol/L, as indicated by continuous glucose monitoring (CGM) readings. Prevention is defined by the avoidance of any CGM interstitial glucose reading below 4.0 mmol/L following the CHO intake. Measured for each intervention visit within 60 minutes after CHO ingestion.

SECONDARY OUTCOMES:
CGM Interstitial Glucose Levels Post-CHO Intake | 10, 15, 20, 30, and 60 minutes
  Continuous glucose monitoring will be used to measure interstitial glucose values at intervals of 10, 15, 20, 30, and 60 minutes after the initial CHO intake. This will assess the glucose response and stability following different CHO dosages and thresholds. Measured post-CHO ingestion during each intervention.
Lowest CGM Glucose Value Post-CHO Intake | 60 minutes
  This outcome will record the lowest CGM glucose reading within 60 minutes following the initial CHO intake for each intervention. This helps determine the effectiveness of the intervention in preventing deep hypoglycemia. Measured within 60 minutes of CHO ingestion during each intervention.
Time Spent in Hypoglycemia Following CHO Intake | 60 minutes
  The duration, in minutes, spent in hypoglycemia (CGM readings < 4.0 mmol/L) within 60 minutes after the initial CHO ingestion will be recorded. This will assess how well each intervention prevents prolonged hypoglycemia. Measured within 60 minutes post-CHO ingestion during each intervention.
Percentage of Episodes Corrected by CHO at Specific Time Intervals | 10, 15, 20, and 30 minutes
  The proportion of hypoglycemic episodes (CGM readings < 4.0 mmol/L) corrected at 10, 15, 20, and 30 minutes after CHO intake will be measured to evaluate the effectiveness of each CHO intervention. Measured at 10, 15, 20, and 30 minutes after CHO ingestion for each intervention.
Number of Episodes Requiring Additional CHO Treatment | 60 minutes
  The number of hypoglycemic episodes that require additional CHO intake after the initial dose will be recorded. This assesses whether the initial CHO intake was sufficient to correct hypoglycemia. Measured within 60 minutes post-CHO ingestion during each intervention.
Incidence of Rebound Hyperglycemia (≥ 10.0 mmol/L) | 60 minutes
  The occurrence of rebound hyperglycemia (CGM reading ≥ 10.0 mmol/L) within 60 minutes following the initial CHO intake will be documented to assess the risk of overcorrection leading to hyperglycemia. Measured within 60 minutes post-CHO ingestion during each intervention.
Total CHO Consumption per Intervention | 60 minutes
  The cumulative amount of CHO consumed per intervention will be recorded to analyze CHO requirements and efficiency across different intervention arms.
Safety Endpoint - Plasma Glucose and CGM Lag-Time Analysis | 5, 10, 15, 20, and 30 minutes
  Plasma glucose levels at specified intervals (5, 10, 15, 20, and 30 minutes after CHO intake) will be compared to CGM readings to assess the lag time between plasma and interstitial glucose during hypoglycemia correction. Measured at 5, 10, 15, 20, and 30 minutes post-CHO ingestion for each intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Remi Rabasa-Lhoret, Principal Investigator — IRCM
Locations (2):
- Canada (2):
  - Institut de recherches cliniques de Montréal, Montreal, Quebec
  - Montreal Clinical Research Institute, Montreal, Quebec